CLINICAL TRIAL: NCT01361503
Title: Magnetic Resonance Spectroscopic and Diffusion Tensor Imaging of Adolescents with Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Instructor in Psychiatry, Massachusetts General Hospital
Other Study IDs: 2010-P-000185
Record Dates: First submitted 2010-11-19; First posted 2011-05-26 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Pervasive Developmental Disorders; Asperger's Syndrome; Adolescents; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder (ASD)
- Controls

SUMMARY:
The primary objective of this study is to conduct magnetic resonance spectroscopic (MRS) and imaging (MRI) scans to assess the structural and neurochemical profile of the brain in 20 children and adolescents, 6-17 years old with Autism Spectrum Disorder (ASD). For comparison, MRS and MRI will also be obtained from 10 healthy control subjects, matched to the 20 subjects with ASD in age, sex, dexterity, and IQ. All eligible subjects will be administered a detailed assessment battery consisting of cognitive assessments (neuropsychological battery including subsets of the DANVA2 and the CANTAB) and measures of psychosocial functioning (SAICA and M-FES). The study includes 1-3 visits for the screening period at Massachusetts General Hospital (approximately 4 hours of assessments) and one scanning visit at McLean Hospital (approximately 1.5 hours).

The investigators hypothesize that youth with ASD versus controls will exhibit increased glutamate concentrations, reflecting glutamatergic overactivity, and increased Cho concentrations, suggesting neuronal abnormality. Furthermore, the investigators hypothesize that compared to neurotypical controls, the structural integrity of white mater tracts will be disrupted in ASD.

ELIGIBILITY:
Inclusion Criteria

* Male or female participants between 6 and 17 years of age.
* Fulfills diagnosis of autism spectrum disorders by meeting DSM-IV-TR PDD diagnostic criteria for autistic disorder, Asperger's disorder, or PDD-NOS as established by clinical interview.
* Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their legal representative must be considered reliable reporters.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative and the subject must sign an IRB approved informed consent and assent document respectively.
* Participants with disruptive behavior disorders, mood and anxiety disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion Criteria

* IQ < 85.
* DSM-IV-TR PDD diagnoses of Rett's disorder, or childhood disintegrative disorder.
* Current diagnosis of a psychotic disorder or unstable bipolar disorder.
* History of recent or current (past 30 days) clinically significant depressive or anxiety disorder that warrants treatment.
* History of substance use (except nicotine or caffeine) within past 3 months or urine drug screen positive for substances of abuse.
* Clinically unstable psychiatric conditions or judged to be at serious safety risk to self (suicidal risk) or others.
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study.
* Organic brain disorders.
* History of non-febrile seizures without a clear and resolved etiology in last 1 month.
* Pregnant or nursing females.
* Left hand dominant subjects.
* History of claustrophobia or fear of enclosed places.
* Presence of metal or surgical devices (aneurysm clips, metal plates, cochlear implants, neurostimulators, braces, and other items).
* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited from current patients of The Alan and Lorraine Bressler Clinic for Autism Spectrum Disorders. We propose to contact by letter (via regular mail or email) or telephone patients who have been identified by clinicians as expressing interest in the study. Subjects who have participated in previous protocols in our program may also be eligible to participate in this study. We propose to contact by letter or telephone past study participants who have expressed interested in being contacted about future studies they may be eligible for in our office. If a potential subject's clinician ascertains that the patient has an interest in study participation, the clinician will only offer contact information for the study to the patient and/or the patient's parents. The patient and/or parent can then contact the study coordinator for more information on the actual study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Structural and neurochemical profiles of adolescents with ASD | scanning visit (1.5 hours)
  Concentrations of various neurochemicals, including glutamate, will be examined in addition to the structural integrity of white matter tracts. These results will be compared to results from control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts